CLINICAL TRIAL: NCT05334420
Title: Efficacy Trial of a Program for Weight Loss for Hispanic Fathers and Increased Physical Activity for Their Children: Healthy Dads, Healthy Kids
Brief Title: Efficacy Trial Healthy Dads, Healthy Kids for Hispanic Fathers and Children
Acronym: HDHK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Newcastle, Australia (Other); San Diego State University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Teresia O'Connor, Professor of Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-50011; R61HL155015 (NIH)
Record Dates: First submitted 2022-04-04; First posted 2022-04-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Obesity, Childhood; Physical Activity; Dietary Intake
Keywords: Hispanic; Latino; Family based intervention; Father
MeSH Terms: conditions — Obesity; Pediatric Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with family unit (minimum of father-child, maximum of father, 3 siblings, and mother/partner) randomized to intervention or standard of care control.
Who Masked: Outcomes Assessor
Masking Description: Staff involved in assessment will be masked to participant allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Dads Healthy Kids (Experimental): A group-based lifestyle behavioral program for Hispanic fathers and children
  Interventions: Behavioral: Healthy Dads Healthy Kids
- Standard of care control (Other): National guidelines and recommendations for healthy eating, physical activity and weight loss.
  Interventions: Other: Standard of care control

INTERVENTIONS:
Behavioral: Healthy Dads Healthy Kids — Group based lifestyle behavioral intervention for weight loss for fathers and increased physical activity for their child. The program meets weekly 90-minute sessions over 10 weeks. Mothers/partners are invited to one session (Week 4). Each meeting consisted of a brief review session with Dads and Kids together (15 minutes), separate break-out discussion for Dads (Dad's Club) and Kids (Kid's Club) (30 minutes); and a joint physical activity component for Dads and Kids (Sports Club) (45 minutes). Each week covers different topics for fathers and a corresponding session for kids. The program encourages fathers to be healthy, positive role models for their children, and teaching fathers weight loss strategies, authoritative parenting strategies and to encourage healthy behaviors in their kids. Fathers and kids are encouraged to eat healthy, reduce their screen time and be more active. If the COVID pandemic prevents in-person meetings, the program will be delivered virtually.
  Other Names: Papás Saludables, Niños Saludables
  Arms: Healthy Dads Healthy Kids
Other: Standard of care control — Families will receive handouts on healthy eating, physical activity and screen media use to promote healthy weight status. Fathers will attend one group session with a focus on dietary changes and increased physical activity to promote healthy weight loss.
  Arms: Standard of care control

SUMMARY:
Hispanic men and children experience health disparities for overweight and obesity-related medical conditions, and therefore family level obesity prevention programs for Hispanic populations are needed. 'Healthy Dads Healthy Kids' is the first program to primarily target fathers for obesity prevention for themselves and their children, with significant and clinically relevant treatment effects. This is an efficacy trial to assess a culturally adapted 'Healthy Dads Healthy Kids' for Hispanic families.

DETAILED DESCRIPTION:
Hispanics in the United States face health disparities for obesity and related medical conditions, such as cardiovascular disease and diabetes. Targeting families to promote healthy lifestyle behaviors has been identified as an effective strategy to prevent obesity. With the importance of familism (family cohesion) among the Hispanic population, a family based intervention is especially desirable as an engaging strategy to promote behaviors that support a healthy weight status and decrease obesity related health disparities for Hispanics. Emerging evidence supports the need to include and target fathers in family based lifestyle behavior interventions. Healthy Dads Healthy Kids (HDHK) is an evidence based program developed in Australia, shown to have significant weight and behavior treatment effects for fathers and their children, compared to controls. The HDHK program is based on Social Cognitive Theory and Family Systems Theory and aims to promote increased physical activity and improved dietary intake for fathers and their children. An important innovation in the program is that fathers and children attend together and are both targeted as agents of behavior change for each other (reciprocal reinforcement) and to participate in fun, family activities together. HDHK was culturally adapted for Hispanic families following the Ecological Validity Model by this research team, with input from a community Hispanic family panel, expert committee and the developer of the HDHK program. The resulting Papás Saludables, Niños Saludables (PSNS) program is a 10-week group-based intervention that meets weekly.

This randomized controlled trial of PSNS is powered to detect a clinically meaningful change in father's weight and children's moderate to vigorous physical activity. The study will also assess other behavioral (dietary intake, sedentary time, screen media use, and parenting practices), psychosocial (familism, acculturation, and co-parenting alliance) and biological (child BMI z-score, father's non-HDL, HgbA1C, and BP) outcomes. Hispanic men with overweight or obesity who are a father figure (biological father, step father, grandfather, adult older brother, etc) to a 5-11 child will be enrolled in the study in waves. Participants are enrolled as a family unit and includes the father, child(ren) (up to 3 siblings) and mother/partner (if available). After screening and baseline data is complete for a wave, the family is randomized to receive a standard of care control or the group-based culturally adapted PSNS. Follow-up assessments will be done at 4 months and 12 months.

The study includes a partnership with the YMCA of Greater Houston to provide a venue for where to deliver the program.

ELIGIBILITY:
FATHER

* Father or significant male role model (e.g. step father, grandfather, uncle, or older brother) of a child 5-11 years old
* Age 18-65 year old
* Living in Greater Houston Area
* Self-identify as Hispanic or Latino
* Able to read and write in Spanish or English
* BMI >/=25 - 40
* Pass the 2015 American College of Sports Medicine's exercise participation health screener

CHILD

• 5-11 year old child and up to three siblings, whose father/significant male role model is participating

MOTHER (If available) 1) Significant female role model such as biological mother, step mother, foster mother, grandmother, aunt or older sister; or other co-parent/partner to participating children

Exclusion Criteria:

FATHER

* Known diagnosis of diabetes without medical clearance from health care provider;
* Known diagnosis of cardio-vascular disease (cardiac arrhythmia, h/o myocardial infarction, heart valve disease, heat failure, heart transplantation, congenital heart disease, h/o heat surgery, coronary angioplasty, or stroke)
* Currently, or in the past 6 months, in a weight management program
* Currently, or in the past 6 months, taking medicine that can affect weight or might be affected by weight loss
* Any other disease or condition affecting their ability to participate in physical activities/exercise (e.g., physical disability, severe asthma)
* Any other disease or condition affecting their ability to participate in group classroom activities including cognitive impairment (e.g., Down's syndrome, Fragile X), or psychiatric functioning (e.g. schizophrenia)
* Plans of moving away from Harris County in the next year
* Not passing the 2015 American College of Sports Medicine's exercise participation health screener AND NOT provide a medical clearance from a licensed medical provider (MD, NNP, PA)
* Unwilling to wear accelerometer for a 7 day study period at the three assessment points.
* BMI less than 25 or greater than 40.
* HbgA1C equal or greater than 6.5% at baseline data collection without medical clearance from health care provider.
* Has previously participated in studies on the Healthy Dads Healthy Kids' for US Hispanics
* History of myocarditis from COVID infection or vaccine

CHILD

* Not within the 5-11 year old child age range
* Known diagnosis of diabetes
* Known diagnosis of cardio-vascular disease (cardiac arrhythmia, h/o myocardial infarction, heart valve disease, heat failure, heart transplantation, congenital heart disease, h/o heat surgery or coronary angioplasty)
* Inability to participate in regular physical education classes in school due to health or physical condition (e.g. physical disability, severe asthma)
* Any disease or condition affecting their ability to participate in group classroom activities including cognitive impairment (e.g. Down's syndrome, Fragile X), or developmental problems (e.g. autism spectrum disorder)
* Any Known diagnosis of an eating disorder (e.g. anorexia nervosa, bulimia nervosa, etc.) MOTHER
* No father figure to her children enrolled in the study

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — In order to participate, a person identified as a child's father figure (male gender) needs to enroll as the target of the study
Enrollment: 187 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Father´s weight | 12 months
  weight in kg
Child´s moderate to vigorous physical activity (MVPA) | 12 months
  MVPA will be measured by Actigraph accelerometer with a minimum of 4 days of data 600 min/day

SECONDARY OUTCOMES:
Father´s weight | 4 months
  weight in kg
Child´s MVPA | 4 months
  MVPA will be measured by Actigraph accelerometer with a minimum of 4 days of data 600 min/day
Father´s MVPA | 4 and 12 months
  MVPA will be measured by Actigraph accelerometer with a minimum of 4 days of data 600 min/day
Child´s and father's dietary intake | 4 and 12 months
  Separate NCI´s ASA 24 hour dietary recalls for dads and kids. One recall at each time-point
Child's BMI z-score | 4 and 12 months
  Height (m) and weight (kg) measured and BMI z score calculated using CDC macro
Child´s and father's screen media use | 4 and 12 months
  Survey of screen use in past week
Father's blood heart rate | 4 and 12 months
  Automatic blood pressure machine
Father's blood pressure | 4 and 12 months
  Automatic blood pressure machine
Fathers's non-HDL | 4 and 12 months
  Cholestech LDX 13-452 Analyzer with the Cholestech LDX; TC/HDL Panel Test Cassette
Father's HgbA1C | 4 and 12 months
  DCA Vantage Analyzer using the DCA Vantage HBA1C test kit
Child's and father's sedentary time | 4 and 12 months
  Sedentary time will be measured by accelerometer with a minimum of 4 days of data 600 min/day
Co-parenting alliance | 4 and 12 months
  Validated survey questionnaire: Co-parenting Alliance Instrument
Father-child bonding | 4 and 12 months
  Validated survey questionnaire: Child-Parent Relationship Scale
Father's food and physical activity parenting practices | 4 and 12 months
  Validated survey questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The principal investigator and co-investigators acknowledge their willingness to share data with other eligible investigators through academically established means. Summarized data will be shared with collaborators as soon as available, with local colleagues at seminars and talks, and with the scientific community at large by posters and presentations at local, regional, national and international scientific meetings.
  Individual participant data may be shared with reasonable requests and data sharing agreements put in place between institutions.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after completion of study (anticipated August 2026)
Access Criteria: Valid research question posed by investigators at an academic institution. IRB approval obtained Data sharing agreement in place

REFERENCES:
- [Background] De Boer RJ, Perelson AS. Towards a general function describing T cell proliferation. J Theor Biol. 1995 Aug 21;175(4):567-76. doi: 10.1006/jtbi.1995.0165. PMID 7475092
- [Background] Godel V, Regenbogen L, Feiler-Ofry V, Lazar M. Vitreoretinal degeneration in facial clefting syndrome. Birth Defects Orig Artic Ser. 1982;18(6):581-6. No abstract available. PMID 7171778
- [Background] Perez O, Beltran A, Isbell T, Galdamez-Calderon E, Baranowski T, Morgan PJ, O'Connor TM. Papas Saludables, Ninos Saludables: Perspectives From Hispanic Parents and Children in a Culturally Adapted Father-Focused Obesity Program. J Nutr Educ Behav. 2021 Mar;53(3):246-253. doi: 10.1016/j.jneb.2020.11.006. Epub 2020 Dec 22. PMID 33358181